CLINICAL TRIAL: NCT01231737
Title: Efficacy of Prulifloxacin vs Phosphomycin in the Prophylasy of Urinary Tract Infection
Brief Title: Efficacy of Two Prophylactic Schedules (Prulifloxacin Versus Phosphomycin)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University Of Perugia (Other)
Responsible Party: University of Perugia, University of Perugia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 002
Record Dates: First submitted 2010-01-14; First posted 2010-11-01 (Estimated); Last update posted 2010-11-01 (Estimated); Status verified 2009-10

CONDITIONS: Urinary Tract Infection
Keywords: Prophylasy; recurrent urinary tract infection; prulifloxacin; phosphomycin
MeSH Terms: conditions — Urinary Tract Infections | interventions — prulifloxacin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Prulifloxacin (Active Comparator)
  Interventions: Drug: prulifloxacin

INTERVENTIONS:
Drug: prulifloxacin — Prulifloxacin 1 tablet/week for 12 weeks.

SUMMARY:
Epidemiological studies showed that 20-30% of patients with uncomplicated urinary tract infections risked recurrent infection. Urinary tract infection causes marked discomfort for the patient, has a negative impact upon quality of life, and is associated with high social and health costs in terms of specialist appointments, laboratory and instrumental tests and prescriptions . Although diverse cycles of antibiotic therapy and prophylaxis have been proposed, doubts persist about the most efficacious pharmacological agents, duration of prophylaxis , the incidence of adverse effects and relapse when antibiotic therapy is suspended.

Aims of the study:

1. To compare the efficacy of two prophylactic schedules (Prulifloxacin vs Phosphomycin):

   * in reducing the number of urinary tract infection episodes during prophylaxis
   * in reducing the number of urinary tract infection episodes after prophylaxis
   * in improving the patient's quality of life .
2. To assess :

   * Tolerability of antibiotic prophylaxis
   * The incidence of resistance to antibiotic therapy

ELIGIBILITY:
Inclusion Criteria:

* Female patients
* Age over 18 years old
* No allergies to the drugs to be prescribed
* No counter-indications to this drug therapy
* Urine culture shows responsiveness to drugs at recruitment of patient
* History of urinary tract infections with at least three episodes in the previous year or two in the past six months

Exclusion Criteria:

* Lack of tolerability of prescribed drugs

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2010-11; Primary Completion 2011-02 (Estimated); Study Completion 2012-02 (Estimated)

PRIMARY OUTCOMES:
number of urinary tract infection episodes during prophylaxis | 3 months

SECONDARY OUTCOMES:
improving the patient's quality of life | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Elisabetta Costantini, Study Chair — University Of Perugia